CLINICAL TRIAL: NCT04545242
Title: Efficacy of Higher vs. Lower Doses of Dexamethasone in Patients With Acute Hypoxemic Respiratory Failure (Including ARDS) Caused by Infections (Including COVID-19)
Brief Title: Efficacy of DEXamethasone in Patients With Acute Hypoxemic REspiratory Failure Caused by INfEctions
Acronym: DEXA-REFINE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Li Ka Shing Knowledge Institute (Unknown); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Jesus Villar, Senior scientist, Dr. Negrin University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICI20-00062
Record Dates: First submitted 2020-09-05; First posted 2020-09-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Acute respiratory failure; ARDS; Mechanical ventilation; Infection
MeSH Terms: conditions — Respiratory Insufficiency; Infections | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled, open-label trial involving mechanically ventilated adult patients with AHRF (including ARDS) caused by confirmed bacterial or viral infections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (low dose) (Active Comparator): Dexamethasone: 6 mg/iv/day during 10 days.
  Interventions: Drug: Dexamethasone
- Dexamethasone (moderate dose) (Active Comparator): Dexamethasone: 20 mg/iv/ daily from day of randomization (day 1) during 5 days, followed by 10 mg/iv/ daily from Day 6 to Day 10 of randomization.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Intravenous dexamethasone (low vs. moderate doses) during 10 days
  Other Names: Decadron; Dexasone; Diodex

SUMMARY:
Background: There are no proven therapies specific for pulmonary dysfunction in patients with acute hypoxemic respiratory failure (AHRF) caused by infections (including Covid-19). The full spectrum of AHRF ranges from mild respiratory tract illness to severe pneumonia, acute respiratory distress syndrome (ARDS), multiorgan failure, and death. The efficacy of corticosteroids in AHRF and ARDS caused by infections remains controversial.

Methods: This is a multicenter, randomized, controlled, open-label clinical trial testing dexamethasone in mechanically ventilated adult patients with established AHRF (including ARDS) caused by confirmed pulmonary or systemic infections, admitted in a network of Spanish ICUs. Eligible patients will be randomly assigned to receive dexamethasone: either 6 mg/d x 10 days or 20 mg/d x 5 days followed by 10 mg/d x 5 days. The primary outcome is 60-day mortality. The secondary outcome is the number of ventilator-free days at 28 days. All analyses will be done according to the intention-to-treat principle.

DETAILED DESCRIPTION:
Acute hypoxemic respiratory failure (AHRF), and its more severe form termed the acute respiratory distress syndrome (ARDS), is a catastrophic illness of multifactorial etiology characterized by a severe inflammatory process of the lung leading to hypoxemic respiratory failure requiring mechanical ventilation (MV). Pulmonary infections are the leading causes of AHRF and ARDS. Translational research has established a strong association between dysregulated systemic and pulmonary inflammation and progression or delayed resolution of AHRF.2 Glucocorticoid receptor-mediated downregulation of systemic and pulmonary inflammation is essential to accelerate disease resolution and restore tissue homeostasis, and can be enhanced with glucocorticoid treatment.

The COVID-19 pandemic is a critical moment for the world, in which even industrially advanced countries have rapidly reached intensive care units (ICUs) saturation, and intensivists are forced to make difficult ethical decisions that are uncommon outside war zones. As with other bacterial or viral infections, severe pneumonia is the main condition leading to AHRF and ARDS requiring weeks of MV with high mortality (35-55%) in critically ill patients. There has been great interest in the role of corticosteroids to attenuate the pulmonary and systemic damage in ARDS patients because of their potent anti-inflammatory and antifibrotic properties.3 Corticosteroids have been off patent for greater than 20 years, they are cheap, and globally equitable. However, the efficacy of corticosteroids in AHRF (including ARDS) caused by infections remains controversial.

Only two large randomized clinical trials (RCT) have shown that the administration of dexamethasone is able to reduce mortality in patients with AHRF. Villar et al in Spain observed that moderate doses of dexamethasone (10-20 mg/d x 10 days) caused a 15% absolute reduction of 60-day mortality in patients with established moderate-to-severe ARDS from multiple etiologies. Horby et al in the RECOVERY trial in Great Britain reported that dexamethasone at low doses (6 mg/d x 10 days) reduced 28-day mortality in patients with AHRF caused by COVID-19. These findings confirmed that corticosteroid therapy is associated with a sizable reduction in duration of MV and hospital mortality. These two RCTs will change clinical practice for the management of AHRF and ARDS. However, there is a reasonable doubt whether dexamethasone at moderate doses (10-20 mg/d) would cause a greater reduction in mortality than 6 mg/d. Our goal in this study is to respond this question.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* intubated and mechanically ventilated;
* acute onset of AHRF (as defined by a PaO2/FiO2 ≤300 mmHg during at least 6 hours from diagnosis. For the measurement of PaO2 and calculation of PaO2/FiO2 ratio, the minimum accepted value for PEEP is 5 cmH2O and for FiO2 is 0.3. ARDS is defined by Berlin criteria,4 which includes: (i) having pneumonia or worsening respiratory symptoms, (ii) bilateral pulmonary infiltrates on chest imaging (x-ray or CT scan), (iii) absence of left atrial hypertension or no clinical signs of left heart failure, and (iv) hypoxemia, as defined by a PaO2/FiO2 ≤300 mmHg on positive end-expiratory pressure (PEEP) of ≥5 cmH2O, regardless of FiO2.
* Pulmonary or systemic infectious etiology of AHRF.

Exclusion Criteria:

* Patients with a known contraindication to corticosteroids,
* Patient included in another therapeutic clinical trial
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
60-day mortality | 60 days
  All-cause mortality at 60 days after randomization

SECONDARY OUTCOMES:
Ventilator-free days | 28 days
  Number of ventilator-free days (VFDs) at Day 28 (defined as days being alive and free from mechanical ventilation at day 28 after randomization. For patients ventilated 28 days or longer and for subjects who die, VFD is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, Principal Investigator — Hospital Universitario Dr. Negrin
Locations (40):
- Spain (40):
  - Hospital Universitario Mutua Terrassa (ICU), Terrassa, Barcelona
  - Hospital General La Mancha Centro (ICU), Alcázar de San Juan, Ciudad Real
  - Complejo Hospitalario Universitario de Santiago (Anesthesia), Santiago de Compostela, La Coruña
  - Hospital General El Bierzo (ICU), Ponferrada, León
  - Hospital Universitario del Henares (ICU), Coslada, Madrid
  - Hospital Universitario de Getafe (ICU), Getafe, Madrid
  - Hospital Universitario Severo Ochoa (ICU), Leganés, Madrid
  - Hospital Universitario Puerta de Hierro (ICU), Majadahonda, Madrid
  - Hospital Nuestra Señora del Prado (ICU), Talavera de la Reina, Toledo
  - Hospital Universitario de Cruces (Anesthesia), Barakaldo, Vizcaya
  - Hospital Universitario de Cruces (ICU), Barakaldo, Vizcaya
  - Hospital Universitario de A Coruña (ICU), A Coruña
  - Complejo Hospitalario Universitario de Albacete (ICU), Albacete
  - Hospital Clinic de Barcelona (AVI), Barcelona
  - Hospital Clinic de Barcelona (Cardiac ICU), Barcelona
  - Hospital Clínic (Hepatic ICU), Barcelona
  - Hospital Clínic de Barcelona (Anesthesia), Barcelona
  - Hospital General de Ciudad Real (ICU), Ciudad Real
  - Hospital Virgen de la Luz (ICU), Cuenca
  - Complejo Asistencial Universitario de León (ICU), León
  - Hospital Universitario La Princesa (ICU), Madrid
  - Hospital Universitario Ramón y Cajal (Anesthesia), Madrid
  - Hospital Clínico Universitario San Carlos (ICU), Madrid
  - Hospital Universitario Fundación Jiménez Díaz (ICU), Madrid
  - Hospital Universitario Doce de Octubre (ICU), Madrid
  - Hospital Universitario La Paz (Anesthesia), Madrid
  - Hospital Universitario La Paz (ICU), Madrid
  - Hospital Universitario Regional de Malaga Carlos Haya (ICU), Málaga
  - Hospital Universitario Virgen de Arrixaca (Anesthesia), Murcia
  - Hospital Universitario Virgen de Arrixaca (ICU), Murcia
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Montecelo (Anesthesia), Pontevedra
  - Hospital Universitario Nuestra Señora de Candelaria (ICU), Santa Cruz de Tenerife
  - Hospital General de Segovia (ICU), Segovia
  - Hospital Clinico Universitario de Valencia (Anesthesia), Valencia
  - Hospital Clinico Universitario de Valencia (ICU), Valencia
  - Hospital Clínico Universitario de Valladolid (Anesthesia), Valladolid
  - Hospital Universitario Río Hortega (Anesthesia), Valladolid
  - Hospital Universitario Río Hortega (ICU), Valladolid
  - Hospital Virgen de la Concha (ICU), Zamora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530